CLINICAL TRIAL: NCT05595070
Title: Oral Complications After Haematopoietic Stem Cell Transplantation: a Retrospective Study
Acronym: RadboudStem
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-13654
Record Dates: First submitted 2022-10-16; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Stem Cell Transplant Complications; Oral Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Haematopoietic stem cell transplantation — Haematopoietic stem cell transplantation (HSCT) is widely used in the treatment of malignant and non-malignant conditions to reconstitute the immune system secondary to cytotoxic conditioning regimens. These regimens, consisting of chemotherapy with or without total body irradiation, cause severe immunosuppression prior to, during and after HSCT. Immune reconstitution takes place by infusion of stem cells either harvested from the patient (autologous HSCT) or from a donor (allogeneic HSCT).

SUMMARY:
Haematopoietic stem cell transplantation (HSCT) is a potentially lifesaving treatment option for various diseases. It involves infusion of stem cells after a conditioning regimen of chemotherapy with or without total body irradiation. There is a concern that HSCT and accompanying treatments may increase the risk for oral complications. Nevertheless, longitudinal studies measuring oral health before and after HSCT are scarce. Hence, we formulated the following research question:

In adult HSCT recipients, do oral health parameters change from baseline (pre-HSCT) to 3 - 24 months post-HSCT, and is the type of conditioning regimen associated with this change in oral health parameters?

To answer this research question, we will use data from the electronic health records of the Radboudumc (Epic and Dentium). We will include at least seventy-five adult patients who are examined both before and after HSCT at the department of Dentistry (Radboudumc) as part of an oral care program. The following oral health parameters were assessed: status praesens, pocket probing depth, bleeding on probing, periodontal epithelial surface area, periodontal inflamed surface area, xerostomia, unstimulated and stimulated salivary flow rate and pH, cariesactivity, oral chronic Graft-versus-Host Disease and dental treatments.

Patients were subjected to different regimens in preparation for HSCT, namely myeloablative, reduced intensity or non-myeloablative conditioning. To estimate the association between conditioning regimen and the change in oral health parameters, we will use mixed effects models with random effects, adjusted for potential confounders. Results will be reported as regression coefficients with corresponding 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic HSCT between 2013 and 2021 at Radboudumc
* Oral focal screening before HSCT, and at least one oral examination after HSCT performed at Department of Dentistry, Radboudumc
* Informed consent

Exclusion Criteria:

* Not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Allogeneic HSCT recipients treated at Radboudumc
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of teeth | Change from baseline (pre-HSCT) up to 24 months after HSCT
  Number of teeth (range 0 - 32)
Number of restorations | Change from baseline (pre-HSCT) up to 24 months after HSCT
  Total number of restored tooth surfaces
Pocket probing depth | Change from baseline (pre-HSCT) up to 24 months after HSCT
  Pocket probing depth at 6 sites per tooth in millimetres
Bleeding on probing | Change from baseline (pre-HSCT) up to 24 months after HSCT
  Profound bleeding on probing at 6 sites per tooth as yes or no
Unstimulated and chewing stimulated salivary flow rate | Change from baseline (pre-HSCT) up to 24 months after HSCT
  Whole mouth saliva, measured in mL/min
Unstimulated and chewing stimulated salivary pH | Change from baseline (pre-HSCT) up to 24 months after HSCT
  Whole mouth saliva, measured with pH strips

SECONDARY OUTCOMES:
Periodontal Epithelial Surface Area | Change from baseline (pre-HSCT) up to 24 months after HSCT
  The root surface area in square millimetres affected by attachment loss
Periodontal Inflamed Surface Area | Change from baseline (pre-HSCT) up to 24 months after HSCT
  The root surface area in square millimetres affected by attachment loss and inflamed periodontal tissue
Xerostomia | Change from baseline (pre-HSCT) up to 24 months after HSCT
  Subjective oral dryness measured by Xerostomia Inventory questionnaire
Cariesactivity | Up to 24 months after HSCT
  Likelihood for development of new caries lesions based on notes recorded by the dentist
Oral chronic Graft-versus-Host Disease | Up to 24 months after HSCT
  Assessed with National Institute of Health Oral Mucosal Score (range 0 - 15), higher score means more severe oral manifestations of oral chronic Graft-versus-Host Disease
Extractions | Between baseline (pre-HSCT) and up to 24 months after HSCT
  Total number of removed teeth (range 0 - 32)
Periodontal care | Between baseline (pre-HSCT) and up to 24 months after HSCT
  Number of participants per type of periodontal care, categorised in sub- and supragingival cleaning, subgingival cleaning, no cleaning
Preventive measures | Between baseline (pre-HSCT) and up to 24 months after HSCT
  Number of participants per type of preventive measure as fluoride varnish and oral hygiene instructions

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided